CLINICAL TRIAL: NCT04313621
Title: Management of Lower Limb Apophysitis: A Cross-sectional Study on Long-term Impact on Health Status
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kasper Krommes, Clinical Research Coordinator, PhD-fellow, Physiotherapist, MSc, Hvidovre University Hospital
Other Study IDs: 123456789
Record Dates: First submitted 2020-03-17; First posted 2020-03-18 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Lower Limb Apophysitis (Severs, Osgood Schlatter, Sinding-Larsen Johansson)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lower limb apophysitis cause long-term pain, decrease in function, and can reduce or completely hinder participation in sports and physical activity, yet there is little knowledge on the long-term consequences for health. Our objective with this investigation is to capture self-reported health-status for all adults having been diagnosed with lower limb apophysitis in the period of 1977 to 2020 and compared these data with normative values for the background population. We are therefore conducting a national cross-sectional study based on data from the Danish National Patient Registry. In this protocol we describe, as detailed as possible, the planned methods.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18-55 having received diagnostics codes pertaining to lower limb apophysitis (Severs, Sinding-Larsen Johansson, Osgood Schlatter) in the years 1977-2020 in Denmark will be eligible to participate.

Exclusion Criteria:

* Diseased participants will be censored

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sample size will be of convenience with no pre-determined cut-off for smallest or largest sample of interest, rather, the final sample of respondents will be based on however many have been designated the diagnostic codes and responds to the survey.
Sampling Method: Non-Probability Sample
Enrollment: 1218 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
Physical and mental health | Baseline
  SF-12 (Short-form 12 item) health survey

SECONDARY OUTCOMES:
Sleep: problems and duration | Baseline
Self-reported level of satisfaction with participation in physical activity and sports | Baseline
  Tegner activity scale (0-10, 10 being no physical activity) and individual specific specific questions
Knee pain | Baseline
  Evaluated on at 0-100 numerical pain rating scale pertaining (0 being no pain) to the knee or other body parts, and worst pain last week or the last month
KOOS subscales | Baseline
  Knee injury and Osteoarthritis Outcome Score (KOOS) and its 5 subscale each scoring 0-100, with 100 being the no problems.
Number of Comorbidities from National Health Survey. and musculoskeletal diagnoses from knee or heel | Baseline
PAS-2 | Baseline
  Physical activtiy scale

CONTACTS AND LOCATIONS:
Locations (1):
- Kasper Krommes, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The full dataset, excluding all personal identifiers, will be posted alongside the pre-print when the results have been disseminated.
Supporting Information: Study Protocol, ICF
Time Frame: After primary publication and for the foreseeable futures thereafter.

REFERENCES:
- [Derived] Krommes K, Bjerre A, Thorborg K, Nielsen MF, Holmich P. Long-Term Knee Health in Adults with a History of Adolescent Osgood-Schlatter: A National Cohort Study of Patients in Secondary Care in Denmark 1977-2020. Sports Med. 2025 Jul;55(7):1769-1781. doi: 10.1007/s40279-025-02214-5. Epub 2025 May 29. PMID 40439870